CLINICAL TRIAL: NCT06646042
Title: A PHASE 1, OPEN-LABEL, FIXED SEQUENCE STUDY TO ESTIMATE THE EFFECT OF CARBAMAZEPINE ON THE PHARMACOKINETICS OF IBUZATRELVIR IN HEALTHY ADULT PARTICIPANTS
Brief Title: A Study to Learn If the Study Medicine Called Carbamazepine Changes How the Body Processes the Other Study Medicine Ibuzatrelvir in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C5091009
Record Dates: First submitted 2024-10-15; First posted 2024-10-17 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: Healthy Participants

STUDY DESIGN:
Intervention Model Description: open-label, 2-period, fixed sequence
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Period 1 (Experimental): ibuzatrelvir single oral dose on Day 1.
  Interventions: Drug: ibuzatrelvir
- Period 2 (Experimental): carbamazepine BID oral doses on Day 1-15. ibuzatrelvir single oral dose on Day 14.
  Interventions: Drug: ibuzatrelvir; Drug: carbamazepine ER

INTERVENTIONS:
Drug: ibuzatrelvir — 2x 300 mg tablet
  Other Names: PF-07817883
Drug: carbamazepine ER — 100 mg BID (Day 1-3) 200 mg BID (Day 4-7) 300 mg BID (Day 8-15)
  Arms: Period 2

SUMMARY:
The purpose of this study is to estimate the effect of carbamazepine, a strong CYP3A4 inducer, on the pharmacokinetics (PK) of ibuzatrelvir in healthy participants.

This study is seeking participants who:

* are male or female that are not of childbearing potential of 18 years of age or older
* are examined to be healthy

The study will consist of two treatments: (1) a single oral dose of ibuzatrelvir 600 mg alone in Period 1 and (2) carbamazepine q12h (BID) titrated from 100 mg to 300 mg over 15 days with a single ibuzatrelvir 600 mg dose coadministered on day 15 in Period 2. All treatments will be taken by mouth.

All participants will remain in the study clinic for 18 days for safety review, laboratory collections, and to collect samples for PK.

All participants selected in the study will be required to go through a screening period up to 28 days. A screening period is the time during which a few participants are examined to see whether they are fit for the study. During this period, the participant's medical history and past and current medications will be reviewed. A series of tests will also be performed to see if they are good to be selected for the study. If the participant meets all required criteria and are interested in continuing, the participant will be brought into the study clinic to stay overnight for 18 days. About 28 to 35 days after discharge following the final treatment, the participant will be contacted for a follow up visit either in person or by telephone. This is to check up on how the participant is doing and to conclude the study.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

-Male participants and female participants who are not of childbearing potential who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, blood pressure, pulse rate and standard 12 lead ECG

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Subjects shown to carry or be positive for HLA-B*1502 or HLA-A*3101 (genotyping alleles/markers related to carbamazepine-associated hypersensitivity reactions, including SJS/TEN).
* Screening supine BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic) for participants <60 years; and ≥150/90 mm/Hg for participants ≥60 years old, following at least 5 minutes of supine rest. If systolic BP is ≥ 140 or 150 mm Hg (based on age) or diastolic ≥90 mm Hg, the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
* An eGFR <60 mL/min/1.73m², as determined by the CKD-EPI equation using Screat calculated using the recommended formulas
* Standard 12-lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, QTcF >450 ms, complete LBBB, signs of an acute or indeterminate- age myocardial infarction, ST-T interval changes suggestive of myocardial ischemia, second- or third- degree AV block, or serious bradyarrhythmias or tachyarrhythmias). If QTcF exceeds 450 ms, or QRS exceeds 120 ms, the ECG should be repeated twice and the average of the 3 QTcF or QRS values used to determine the participant's eligibility. Computer-interpreted ECGs should be overread by a physician experienced in reading ECGs before excluding a participant.
* Participants with ANY of the following abnormalities in clinical laboratory tests at screening and prior to dosing in each period, as assessed by the study-specific laboratory and confirmed by a single repeat test, if deemed necessary: ALT, AST, Bilirubin ≥1.5 x ULN. Participants with an elevated total bilirubin consistent with Gilberts Disease may have a direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ ULN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-10-28 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2025-01-17 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of ibuzatrelvir | Hour 0, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48 post-dose in each period
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) of ibuzatrelvir | Hour 0, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48 post-dose in each period
  if data permits
Area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration (AUClast) ofibuzatrelvir | Hour 0, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48 post-dose in each period

SECONDARY OUTCOMES:
Number of Participants With Treatment Emergent Treatment-Related Adverse Events (AEs) | Baseline (Day 0) up to 35 days after last dose of study medication
Number of Participants With Clinically Significant Change From Baseline in Laboratory Abnormalities | Baseline up to Day 18
Number of Participants With Clinically Significant Change From Baseline in Vital Signs | Baseline up to Day 18

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - New Haven, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5091009